CLINICAL TRIAL: NCT01581073
Title: Prevention of End Stage Kidney Disease by Darbepoetin Alfa In CKD Patients With Non-diabetic Kidney Disease
Brief Title: PRevention of End Stage Kidney Disease by Darbepoetin Alfa In Chronic Kidney Disease Patients With nondiabeTic Kidney Disease
Acronym: PREDICT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Showa University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIGU1115; UMIN000006616 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Chronic Kidney Disease; Diabetes
Keywords: renal anemia; erythropoiesis stimulating agent; hemoglobin; non-diabetes; CKD; Chronic Kidney Disease patients without diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Darbepoetin alfa

ARMS (2):
- High Hb group (Experimental): Darbepoetin alfa is given to the patients. Target Hb level is 12.0g/dL and it should be maintained greater than or equal to 11.0g/dL and less than 13.0g/dL. If the patients do not have medical history of myocardial infarction, stroke, pulmonary embolism, unstable angina, or peripheral artery disease, the target Hb level will be greater than or equal to 12.0g/dL and less than 13.0g/dL. Maximum dose of darbepoetin alfa is 240 microgram per 4 weeks.
  Interventions: Drug: Darbepoetin alfa
- Low Hb group (Active Comparator): Darbepoetin alfa is given to the patients. Target Hb level is 10.0g/dL and it should be maintained greater than or equal to 9.0g/dL and less than 11.0g/dL. If the Hb level exceeds 10.0g/dL in patients, reduce the dose amount or stop giving dose.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Darbepoetin alfa is used for targeting Hb level of 11-13g/dL in high Hb group, and 9-11g/dL in low Hb group.

SUMMARY:
The purpose of this study is to ask whether treating non-diabetic chronic kidney disease (CKD) patients with GFR 8-20mL/min/1.73m2 by darbepoetin Alfa targeting Hb between 11.0 and 13.0g/dL preserves renal function better than targeting Hb between 9.0 and11.0g/dL. The investigators also ask whether the higher Hb targeting 11 to 13g/dL will not cause higher adverse events regarding cardiovascular diseases compared with lower Hb targeting 9 to 11g/dL.

DETAILED DESCRIPTION:
Anemia is common among patients with chronic kidney disease (CKD) and is associated with an increased risk of cardiovascular and renal events. Although erythropoiesis stimulating agent (ESA) has been used to correct anemia, use of ESA (hemoglobin level at approximately 13 g/dL) did not reduce cardiovascular or renal events in diabetic CKD patients. Subgroup analysis of a recent randomized study suggested that use of darbepoetin alfa targeting Hb between 11 and 13 g/dL may preserve renal function better than targeting Hb between 9 and 11g/dL in non-diabetic CKD patients.

ELIGIBILITY:
Inclusion Criteria:

1. CKD patients who have not received chronic dialysis
2. eGFR 8 and more and less than 20 mL/min/1.73m2 determined twice in last 12 weeks.
3. CKD patients with renal anemia at Hb less than 10g/dL within last 8 weeks
4. CKD patients with TSAT 20% and higher or serum ferritin 100ng/mL and higher.
5. CKD patients treated with standard care
6. CKD patients provided written informed consent.

Exclusion Criteria:

1. Diabetes (treated, or HbA1c 6.4% IFCC)
2. CKD patients treated with ESA other than epoetins and darbepoetin.
3. CKD patients treated with epoetin 24000 IU/4w or more.
4. CKD patients treated with darbepoetin 90μg/4w or more.
5. Uncontrolled hypertension (180/10mmHg and higher)
6. Heart failure (NYHA III and IV)
7. malignancy, hematological disorder
8. malnutrition
9. Active and continuous gastrointestinal tract bleeding
10. ANCA associated glomerulonephritis, acute infection, active SLE
11. CKD patients who will undergo dialysis or receive transplantation within 6 months
12. Myocardial infarction within last 6 months
13. Stroke or pulmonary embolism within last 12 months
14. Severe allergy
15. Pregnant women, women on lactation, or CKD patients who plant to get pregnant
16. Allergy against erythropoetin
17. Ineligible patients according to the investigator's judgment

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2012-02-16 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Composite renal outcome of chronic dialysis, kidney transplantation, eGFR 6 mL/min/1.73m2 or less, or eGFR less than 50% of initial value. | 96 weeks

SECONDARY OUTCOMES:
Composite cardiovascular outcome of cardiovascular death, stroke, myocardial infarction, leg amputation, admission by heart failure or angina. | 96 weeks
Time from enrollment to initiation of dialysis | 96 weeks
Time from enrollment to 50% reduction of eGFR from initial value | 96 weeks
Time from enrollment to death by any cause | 96 weeks
Change of eGFR from enrollment | 96 weeks
Change of proteinuria/Cr ratio | 96 weeks
Renal protection in patients who maintained the target Hb more than half the time | 96 weeks
50% renal survival | 96 weeks
Stroke | 96 weeks
Myocardial infarction | 96 weeks
Development of malignancy | 96 weeks
Number of Participants with Adverse Events baseline | 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Showa University School of Medicine, Shinagawa, Tokyo, Japan

REFERENCES:
- [Derived] Maruyama S, Kurasawa S, Hayashi T, Nangaku M, Narita I, Hirakata H, Tanabe K, Morita S, Tsubakihara Y, Imai E, Akizawa T; PREDICT Investigators. Higher hemoglobin levels using darbepoetin alfa and kidney outcomes in advanced chronic kidney disease without diabetes: a prespecified secondary analysis of the PREDICT trial. Clin Exp Nephrol. 2023 Sep;27(9):757-766. doi: 10.1007/s10157-023-02362-w. Epub 2023 Jun 8. PMID 37289335
- [Derived] Hayashi T, Maruyama S, Nangaku M, Narita I, Hirakata H, Tanabe K, Morita S, Tsubakihara Y, Imai E, Akizawa T; PREDICT Investigators. Darbepoetin Alfa in Patients with Advanced CKD without Diabetes: Randomized, Controlled Trial. Clin J Am Soc Nephrol. 2020 May 7;15(5):608-615. doi: 10.2215/CJN.08900719. Epub 2020 Apr 3. PMID 32245781
- [Derived] Imai E, Maruyama S, Nangaku M, Hirakata H, Hayashi T, Narita I, Kono H, Nakatani E, Morita S, Tsubakihara Y, Akizawa T. Rationale and study design of a randomized controlled trial to assess the effects of maintaining hemoglobin levels using darbepoetin alfa on prevention of development of end-stage kidney disease in non-diabetic CKD patients (PREDICT Trial). Clin Exp Nephrol. 2016 Feb;20(1):71-6. doi: 10.1007/s10157-015-1133-z. Epub 2015 Jun 17. PMID 26081567